CLINICAL TRIAL: NCT02223507
Title: A Single-blind, Placebo-controlled Single Dose Tolerance Study in Healthy Elderly Male and Female Volunteers After Intravenous Administration of BIIR 561 CL as Loading Dose (Dosage: 75 mg/h, Infusion Time 1 Hour) Followed by Maintenance Dose (Dosage: 40 mg/h and 75 mg/h, Infusion Time 5 Hours)
Brief Title: Single Dose Followed by Maintenance Dose Tolerance Study of BIIR 561 CL in Healthy Elderly Male and Female Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 600.6
Record Dates: First submitted 2014-08-21; First posted 2014-08-22 (Estimated); Last update posted 2014-08-22 (Estimated); Status verified 2014-08

CONDITIONS: Healthy
MeSH Terms: interventions — irampanel

ARMS (2):
- BIIR 561 CL (Experimental)
  Interventions: Drug: BIIR 561 CL
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BIIR 561 CL
  Arms: BIIR 561 CL
Drug: Placebo
  Arms: Placebo

SUMMARY:
The objective of the present study was to obtain information about the safety, tolerability and pharmacokinetics of BIIR 561 CL after continuous intravenous administration of two increasing doses in healthy elderly volunteers, following the infusion schema of a loading dose (1 hour) and a maintenance dose (5 hours)

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female volunteers
* Age >= 60 years
* Broca index from -25% to +25%
* Written informed consent prior to admission to the study

Exclusion Criteria:

* Any finding of the medical examination (including blood pressure, pulse rate and Electrocardiogram (ECG)) deviating from normal and of clinical relevance
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders (exclusion: substitution therapy regarding thyroid gland and/or ovaries)
* Diseases of the central nervous system (CNS) (such as epilepsy) or psychiatric disorders or neurological disorders and medical history of such diseases or disorders
* History of orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* Allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* Intake of drugs with a long half-life (> 24 hours) within at least one month or less than ten half-lives of the respective drug before enrolment in the study
* Intake of any drugs which might influence the results of the trial (<= one week prior to administration or during the trial)
* Participation in another trial with an investigational drug (<= two months prior to administration or during the trial
* Smoker (> 10 cigarettes or > 3 cigars or > 3 pipes/day)
* Inability to refrain from smoking on trial days
* Alcohol abuse (> 30g/day for males, > 24 g for females)
* Drug abuse
* Blood donation (>= 100 ml within four weeks prior to administration or during the trial)
* Excessive physical activities (within the last week before the study)
* Any laboratory value outside the reference range of clinical relevance

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13
Dates: Start 2000-08; Primary Completion 2000-09 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events | up to 8 days after drug administration
Number of subjects with clinically significant findings in vital functions | up to 8 days after drug administration
  blood pressure, pulse rate, respiratory rate, oral body temperature
Number of subjects with clinically significant findings in ECG | up to 8 days after drug administration
Number of subjects with clinically significant findings in laboratory tests | up to 8 days after drug administration

SECONDARY OUTCOMES:
Maximum drug plasma concentration (Cmax) | up to 32 hours after first drug administration
Time to Cmax (tmax) | up to 32 hours after first drug administration
Terminal half-life (t1/2) | up to 32 hours after first drug administration
Area under the plasma concentration-time curve from zero to the last time points with a quantifiable plasma concentration (AUC0-tf) | up to 32 hours after first drug administration
Area under the plasma concentration-time curve extrapolated to infinity (AUC0-inf) | up to 32 hours after first drug administration
Mean residence time (MRT) | up to 32 hours after first drug administration
Plasma clearance (CL) | up to 32 hours after first drug administration
Volume of distribution (Vz) | up to 32 hours after first drug administration
Volume of distribution at steady state (Vss) | up to 32 hours after first drug administration
Amount excreted into urine (Ae) | up to 32 hours after first drug administration